CLINICAL TRIAL: NCT00720330
Title: The Effect of Thoracolumbar Paravertebral Block or Intravenous Lidocaine and Ketamine Versus Standard Care on Acute and Chronic Pain After Inguinal Herniorrhaphy
Brief Title: Lidocaine and Ketamine Versus Standard Care on Acute and Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment challenges prohibited study progression.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kenneth Cummings III, MD, MS, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-385
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Pain; Nausea
Keywords: Inguinal Herniorrhaphy; Pain assessment; Outcomes
MeSH Terms: conditions — Pain; Nausea | interventions — Ropivacaine; Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine (Active Comparator): Paravertebral Group - A local anesthetic (ropivacaine) will be injected near the spine before surgery. Participants will also receive midazolam and fentanyl intravenously (through your vein) for sedation
  Interventions: Drug: ropivacaine
- Lidocaine/ketamine (Active Comparator): Participant will receive general anesthesia through the vein before surgery. Lidocaine and ketamine will be administered intravenously throughout surgery and for 60 minutes after surgery.
  Interventions: Drug: Lidocaine/Ketamine
- Placebo (Placebo Comparator): General anesthesia plus placebo. Placebo will be administered intravenously until 60 minutes after surgery
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ropivacaine — 10 ml 0.5% ropivacaine plus epinephrine will be injected at T11 and L1 as described above (20 ml total) using intravenous midazolam (1-2 mg) and fentanyl (0.5-1 mcg/kg) for sedation
  Arms: Ropivacaine
Drug: Lidocaine/Ketamine — Patients will receive a general anesthetic consisting of intravenous induction with lidocaine (1.5 mg/kg), propofol (1.5-2.5 mg/kg), ketamine (0.25 mg/kg), fentanyl (1 mcg/kg), and midazolam (1-2 mg).
  Arms: Lidocaine/ketamine
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
The investigators are conducting this study to find out if intravenous (injected through the vein) infusion of lidocaine and ketamine administered with general anesthesia is as effective as a paravertebral block in lessening pain after surgery and that both of these techniques are superior to general anesthesia alone in reducing pain immediately after surgery and in the long-term.

DETAILED DESCRIPTION:
Participants will be randomized into one of three study groups; Group 1 - Paravertebral Group - ropivacaine is injected near the spine before surgery. Midazolam and fentanyl are administered intravenously for sedation. Group 2 - Lidocaine/Ketamine - General anesthesia with lidocaine and ketamine administered intravenously throughout your surgery and for 60 minutes after surgery. Group 3 - General Anesthesia Alone. General anesthesia with placebo administered intravenously throughout surgery and for 60 minutes after surgery. All participants will rate their pain on a scale from 0 to 10 after surgery and on days 1 and 2 after surgery. Participants are called 3 and 6 months after surgery for pain and quality of life assessments

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 75 years
* Male
* Unilateral inguinal hernia scheduled for elective open repair

Exclusion Criteria:

* Incarcerated hernia or urgent procedure
* Reoperation (recurrent hernia)
* Contraindication to regional anesthesia such as:
* Coagulopathy
* Infection at the site of needle insertion
* Pre-existing chronic pain (at any site) requiring treatment
* Contraindication to any study medication (local anesthetic or ketamine)
* History of significant Axis I psychiatric disease (major depressive disorder,bipolar disorder, schizophrenia, etc.)
* Significant hepatic (ALT or AST > 2 times normal) or renal (serum creatinine > 2 mg/dl) impairment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cummings, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic/Hillcrest Hospital, Mayfield Heights, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
Started | 5 | 4 | 3
Completed | 5 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12) | 52 (10) | 53 (13) | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 4 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 5 | 4 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 90 (13) | 77 (14) | 101 (13) | 88 (15)
Height [Mean (Standard Deviation); unit: cm] | 176 (10) | 183 (5) | 179 (13) | 179 (7)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Consumption in Oral Oxycodone Equivalents
Description: The cumulative opioid consumption after surgery until the end of second postoperative day.
Time Frame: 2 days after surgery
Measure: Mean (Full Range); unit: mg
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
Number analyzed (Participants) | 5 | 4 | 3
mg | 564 [0 to 2645] | 73 [30 to 170] | 1381 [25 to 2450]

2. Secondary Outcome: Pre- and Intra-operative Opioid Consumption in Fentanyl Equivalents
Description: The cumulative opioid consumption is calculated as fentanyl equivalent
Time Frame: From admission to the end of surgery
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
Number analyzed (Participants) | 5 | 4 | 3
mcg | 100 (50) | 113 (25) | 134 (58)

3. Secondary Outcome: Time From the End of Surgery to Readiness for Hospital Discharge.
Time Frame: Until hospital discharge, assessed up to 6 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
Number analyzed (Participants) | 5 | 4 | 3
hours | 2.2 (0.3) | 3.8 (1.0) | 3.0 (0.3)

4. Secondary Outcome: Pain Scores on Numerical Rating Scale
Description: Numerical Rating Scales is a measurement of pain ranging from 0 to 10 (11 point scale), where 0 is equal to no pain and 10 is equal to worst possible pain. Pain scores were measured in PACU, first and second postoperative mornings.
Time Frame: After surgery until the second postoperative mornings.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
Number analyzed (Participants) | 5 | 4 | 3
units on a scale
  PACU | 0.8 (1.8) | 2.0 (4.0) | 6.3 (1.5)
  POD1 | 4.6 (1.9) | 3.3 (1.9) | 3.7 (2.1)
  POD2 | 2.6 (0.5) | 2.8 (1.3) | 2 (1.0)

5. Secondary Outcome: Postoperative Nausea
Description: Number of patients who had postoperative nausea or vomiting were recorded.
Time Frame: After surgery until the second postoperative day.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
Number analyzed (Participants) | 5 | 4 | 3
Participants | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ropivacaine | Lidocaine/Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes